CLINICAL TRIAL: NCT06205186
Title: Four Pillars of Defense: A Whole Health Approach to the Military
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Tiffany Stewart, Professor, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PBRC 2023-073
Record Dates: First submitted 2023-12-19; First posted 2024-01-12 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Health Behavior
Keywords: Soldier; Resilience
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Program Users (Other)
  Interventions: Behavioral: Army Health

INTERVENTIONS:
Behavioral: Army Health — A whole health mobile application for Soldiers

SUMMARY:
The overall objectives of this study are to better define the construct of psychological resilience in the military, to identify potential modifiable risk factors and trainable skills of psychological resilience in Soldiers, and provide a scalable, integrated physical and mental optimization training app to be integrated into relevant systems. The proposed work would be a first step in identifying predictive risk factors that can be modified to increase the future resilience of Soldiers. With this crucial information, the investigators aim to gather data that will inform the development of a resilience-focused intervention (e.g., a skills training program) and test the feasibility of that intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 21+ and either a Soldier in the NG or NG family member

Exclusion Criteria:

* Under age 21 and not an NG Soldier or family member

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Resilience | 1 month
  Connor Davidson Resilience Scale (CDRISC)
Resilience | 1 month
  Brief Resilience Scale (BRS)
Emotion Regulation | 1 month
  Difficulty in Emotion Regulation Scale (DERS)
Experiential Avoidance | 1 month
  Multidimensional Experiential Avoidance Questionnaire (MEAQ-30)
Intolerance of Uncertainty | 1 month
  Intolerance of Uncertainty Scale (IUS-12)
Coping | 1 month
  Brief COPE
Positive and Negative Social Exchanges | 1 month
  Positive and Negative Social Exchanges (PANSE)
Post Traumatic Stress Disorder (PTSD) | 1 month
  PTSD Checklist (PCL-5)
Sleep | 1 month
  Pittsburgh Sleep Quality Index (PSQI)
Social Support | 1 month
  Social Support Survey (SSS)
Responses to Stressful Experiences | 1 month
  Responses to Stressful Experiences Scale (RSES)
Unit Cohesion | 1 month
  Questionnaire
Depression | 2 weeks
  Patient Health Questionnaire (PHQ-8)
Anxiety | 2 weeks
  Generalized Anxiety Disorder (GAD7)
Stress | 1 month
  Perceived Stress Scale (PSS)
Drug Abuse | 12 months
  Drug Abuse Screening Test (DAST-10)

SECONDARY OUTCOMES:
Topics Ranking | 1 month
  Questionnaire
Technology Use | 1 month
  Questionnaire
Program Satisfaction | 6 Months
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No